CLINICAL TRIAL: NCT07235917
Title: A Phase 2, Double-Blind, Placebo-Controlled Study to Investigate the Safety and Efficacy of Mibavademab in Adult Women With Functional Hypothalamic Amenorrhea
Brief Title: A Study to Investigate Mibavademab in Adult Women With Functional Hypothalamic Amenorrhea
Acronym: KYRIAD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R4461-FHA-2485
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Functional Hypothalamic Amenorrhea (FHA)
Keywords: Secondary amenorrhea; Hypothalamic-Pituitary-Ovarian (HPO) axis; Group I ovulation disorder; Hypogonadotropic hypogonadal anovulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mibavademab (Experimental)
  Interventions: Drug: Mibavademab
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Mibavademab — Administered per the protocol
  Other Names: REGN4461
  Arms: Mibavademab
Other: Placebo — Administered per the protocol
  Arms: Placebo

SUMMARY:
This study is researching an experimental drug called mibavademab (also called "study drug"). The study is focused on patients with a condition called Functional Hypothalamic Amenorrhea (FHA). FHA is a condition where a woman stops menstruating because the brain is not sending the correct hormonal signals to the ovaries, which then are not able to cycle and ovulate properly.

The aim of the study is to see how well the study drug helps the body make the hormones necessary for ovulation and reproduction, and to assess its safety.

The study is looking at several other research questions, including:

* Whether the drug helps bone health
* What side effects may happen from taking the study drug
* How much study drug is in the blood at different times
* Whether the body makes antibodies against the study drug (which could make the drug less effective or could lead to side effects)

ELIGIBILITY:
Key Inclusion Criteria:

1. Diagnosis of FHA after exclusion of anatomic or organic causes of amenorrhea
2. Has had no menstrual bleeding episode within 3 months (or longer) prior to day 1, as described in the protocol
3. Has a Body Mass Index (BMI) ≥18.5 and <25 kg/m^2 at screening, or BMI ≥25 to <30 kg/m^2 at screening AND percentage of body fat <20% from rigorous exercise as determined by the investigator through Standard of Care (SoC) methods (eg, skinfold thickness, DXA, bioimpedance) within 6 months of screening, as described in the protocol

Key Exclusion Criteria:

1. Has presence of primary amenorrhea (failure to reach menarche, first menstrual cycle)
2. Has blood estradiol ≥50 pg/mL or blood progesterone ≥1 ng/mL at screening
3. Has uterine (eg, absence of uterus, prior endometrial ablation, endometriosis, outflow tract disorders) or ovarian (eg, absence of an ovary, presence of polycystic ovaries) conditions that impact assessment of menses or of the HPO axis
4. Has conditions other than FHA that may cause amenorrhea or menstrual cycle disturbances (eg, polycystic ovarian syndrome, hyperprolactinemia, primary ovarian insufficiency, untreated primary hypothyroidism, primary hyperthyroidism)
5. Polycystic ovarian morphology with an ovarian volume >10 cc on TransVaginal UltraSound (TVUS) [or TransAbdominal Pelvic Ultrasound (TAPU) if applicable] at baseline
6. Presence of follicle ≥17 mm, evidence of ruptured follicle, and/or evidence of corpus luteum on TVUS (or TAPU if applicable) at baseline

NOTE: Other protocol-defined Inclusion/Exclusion criteria apply

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 34 (Estimated)
Dates: Start 2026-02-06 (Estimated); Primary Completion 2027-08-23 (Estimated); Study Completion 2027-12-08 (Estimated)

PRIMARY OUTCOMES:
Change from the highest serum estradiol observed during a 28-day period | Baseline to month 6

SECONDARY OUTCOMES:
Change from the mean serum estradiol observed during a 28-day period | Baseline to month 6
Occurrence of menses followed by mid-cycle serum estradiol ≥200 pg/ml and mid-luteal serum progesterone ≥7.9 ng/ml | At month 6
Change in the highest serum estradiol | Baseline through 6 months
Occurrence of serum estradiol ≥200 pg/ml | Through 6 months
Number of ovulatory menstrual cycles | Through 6 months
Number of menses with mid-luteal serum progesterone ≥7.9 ng/ml and midluteal estradiol ≥100 pg/ml | Through 6 months
Number of menstrual cycles | Through 6 months
Percent change in Bone Mineral Density (BMD) at the lumbar spine, as measured by Dual X-ray Absorptiometry (DXA) | Baseline to 6 months
Absolute change in BMD at the lumbar spine, as measured by DXA | Baseline to 6 months
Percent change in Bone Mineral Content (BMC) at the lumbar spine, as measured by DXA | Baseline to 6 months
Absolute change in BMC at the lumbar spine, as measured by DXA | Baseline to 6 months
Percent change in BMD at the lumbar spine, as measured by DXA in participants with baseline lumbar spine BMD Z-score <-1 | Baseline to 6 months
Absolute change in BMD at the lumbar spine, as measured by DXA, in participants with baseline lumbar spine BMD Z-score <-1 | Baseline to 6 months
Percent change in BMC at the lumbar spine, as measured by DXA, in participants with baseline lumbar spine BMD Z-score <-1 | Baseline to 6 months
Absolute change in BMC at the lumbar spine, as measured by DXA, in participants with baseline lumbar spine BMD Z-score <-1 | Baseline to 6 months
Occurrence of Treatment Emergent of Adverse Events (TEAEs) | Up to day 280
Severity of TEAEs | Up to day 280
Concentrations of total mibavademab in serum | Up to day 280
Occurrence of Anti-Drug Antibodies (ADA) to mibavademab | Up to day 280
Magnitude of ADA to mibavademab | Up to day 280

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (2):
- United States (2):
  - Zillan Clinical Research, Houston, Texas
  - Tidewater Clinical Research - Tidewater Physicians for Women, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/